CLINICAL TRIAL: NCT03608462
Title: Modulation of rTMS on Hippocampal Neurogenesis and Functional Network in Early Schizophrenia
Brief Title: Modulation of Repetitive Transcranial Magnetic Stimulation on Hippocampal Neurogenesis and Functional Network in Patients With Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YG2017ZD13
Record Dates: First submitted 2018-07-09; First posted 2018-08-01 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-01

CONDITIONS: Schizophrenia
Keywords: first episode schizophrenia; rTMS; hippocampal neurogenesis; MRS; cognitive function
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Intervention Model Description: In this research,we combine a cross-sectional case control study and a randomized controlled study.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- rTMS targeting the right DLPFC (Sham Comparator): 60 patients will be randomly allocated into this group,half of them will receive iTBS on the right DLPFC,while the other half will receive sham stimulation.
  Interventions: Device: repetitive transcranial magnetic stimulation(DLPFC)
- rTMS targeting the left LPC (Sham Comparator): 60 patients will be randomly allocated into this group,half of them will receive iTBS on left LPC,while the other half will receive sham stimulation.
  Interventions: Device: repetitive transcranial magnetic stimulation(LPC)
- Observation group (No Intervention): To investigate the abnormalities of hippocampal neurogenesis in patients with early schizophrenia(n=30) compared to healthy controls(n=30)

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation(DLPFC) — high frequency(20Hz) repetitive transcranial magnetic stimulation on dorsolateral prefrontal cortex(DLPFC) .Duration:10 days.
  Arms: rTMS targeting the right DLPFC
Device: repetitive transcranial magnetic stimulation(LPC) — high frequency(20Hz) repetitive transcranial magnetic stimulation on left parietal cortex(LPC).Duration:10 days
  Arms: rTMS targeting the left LPC

SUMMARY:
Based on the hypothesis that high-frequency repetitive transcranial magnetic stimulation(rTMS) on the right dorsolateral prefrontal cortex(DLPFC) and left parietal cortex(LPC) could normalise cognitive abnormalities by promoting hippocampal neurogenesis and cortical-hippocampal function in patients with schizophrenia,this research plan to utilise multimodal functional magnetic imaging method(including structural MRI,resting-state functional magnetic resonance imaging and 1H-MRS) to investigate therapeutic efficacy of intermittent theta burst stimulation (iTBS) on cognitive impairment in SZ patients with memory defects,as well as to elucidate the correlation between treatment effects and hippocampal neuroplasticity.

DETAILED DESCRIPTION:
This study includes 150 schizophrenia patients and 30 healthy controls.This study will investigate 1).abnormalities of hippocampal neurogenesis in patients with schizophrenia compared to healthy controls by using 1H-MRS technique 2a).potential modulation effects of repetitive transcranial magnetic stimulation(rTMS) on hippocampal neurogenesis and cortical-hippocampal function of patients with schizophrenia 2b).the optimal rTMS therapy pattern on promoting hippocampal neurogenesis and improving cortico-hippocampal function by comparing the outcome of stimulating two regions(right dorsolateral prefrontal cortex or left parietal cortex) respectively 3).the therapeutic efficacy of rTMS on cognitive impairments and other psychotic symptoms of patients with schizophrenia by adopting cognitive function and psychotic symptoms evaluation,as well as to explore the optimal rTMS treatment pattern on cognitive function by comparing the outcome of stimulating two regions(DLPFC or LPC) respectively 4)association between therapeutic efficacy of rTMS on cognitive deficits and rTMS modulation on hippocampal neurogenesis and its network function,in order to elucidate the underlying mechanism of therapeutic effects of rTMS on cognitive dysfunction in schizophrenia.

ELIGIBILITY:
* Early schizophrenia group:

Inclusion Criteria:

1. The Structured Interview for Prodromal Symptoms (SIPS) was employed.
2. Meet the diagnostic criteria of Diagnostic and Statistical Manual Diploma in Social Medicine(DSM-V) schizophrenia or schizophreniform psychosis.
3. 18-50years of age,right-handed,normal vision or corrected vision, Han nationality.
4. Disease course less than 5 years.
5. Written informed consent

Observation group: First-episode, In addition to criteria1-3,5,antipsychotics naïve,or antipsychotics withdrawal for more than 3 months.

Intervention group:In addition to criteria 1-6,currently under medication and medically stable for at least 1 month(PANSS score fluctuation<10%);continue the original antipsychotics for at least 1 months after recruitment,with consent of the patients,their psychiatrists and family members.

Exclusion criteria:

Current or past neurological illness,severe physical illness,substance abuse or addiction,alcohol dependence,mental retardation,pregnancy or lactation,extreme agitation, stupor, negative suicide,or those who can not cooperate.A history of MECT within 6 months,or those with contraindications to MRI,rTMS.Medically unstable for at least 1 month (PANSS score fluctuation>10%)

* Healthy controls:

Inclusion Criteria:

1. The Structured Interview for Prodromal Symptoms (SIPS) was employed
2. Matched to the early schizophrenia group in terms of age,sex ratio,handedness,and estimated premorbid IQ
3. normal vision or corrected vision, Han nationality
4. Written informed consent

Exclusion Criteria:

History of psychiatric disease in the subjects themselves or a family history of mental disorder in their first-degree relatives,neurological illness,severe physical illness,substance abuse or alcohol dependence,mental retardation.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in MATRICS Consensus Cognitive Battery | baseline,24 hours after the rTMS treatment,30 days
  MATRICS Consensus Cognitive Battery
Change of hippocampal neurogenesis(from baseline) | baseline,24 hours after the rTMS treatment
  Quantify neural stem cells in hippocampal by using H1-MRS
Change of cortical-hippocampal functional network(from baseline) | baseline,24 hours after the rTMS treatment
  Resting-state fMRI data are acquired
Change from baseline in associative memory | baseline,24 hours after the rTMS treatment,30 days
  associative memory

SECONDARY OUTCOMES:
Change from baseline in Positive and Negative Syndrome Scale(PANSS) | baseline,24 hours after the rTMS treatment,30 days
  Positive and Negative Syndrome Scale(PANSS)
Change from baseline in the Scale for the Assessment of Negative Symptoms(SANS) | baseline,24 hours after the rTMS treatment,30 days
  Scale for the Assessment of Negative Symptoms
Change from baseline in UCSD Performance-based Skills Assessment-Brief(UPSA-B) | baseline,24 hours after the rTMS treatment,30 days
  UCSD Performance-based Skills Assessment-Brief

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Mental Health Center, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li X, Xiang Q, Cen H, Zhai Z, Gao T, Lu C, Dong Y, Ye Y, Zhang C, Zhuo K, Wang Y, Liu D. Efficacy of Cortical-Hippocampal Target Intermittent Theta Burst Stimulation (iTBS) on Associative Memory of Schizophrenia: A Double-Blind, Randomized Sham-Controlled Trial. Neuropsychiatr Dis Treat. 2024 Oct 10;20:1941-1955. doi: 10.2147/NDT.S468219. eCollection 2024. PMID 39411184